CLINICAL TRIAL: NCT04380415
Title: Fitbit Atrial Fibrillation From PPG Data Validation Study
Brief Title: Validation of Software for Assessment of Atrial Fibrillation From PPG Data Acquired by a Wearable Smartwatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fitbit LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 129-0469-01
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Detection Notification (Active Comparator): Pulse rate data will be collected from a commercial device worn on the wrist. ECG will be collected from a single lead ambulatory ECG patch worn on the chest. The data from both the commercial wrist-worn device and the ECG patch are not analyzed real-time.
  Interventions: Diagnostic Test: Single lead ambulatory ECG patch
- Non Detection Notification (No Intervention): Pulse rate data will be collected from a commercial device worn on the wrist.

INTERVENTIONS:
Diagnostic Test: Single lead ambulatory ECG patch — Single lead ambulatory ECG patch worn on the chest
  Arms: Detection Notification

SUMMARY:
Validate the Fitbit PPG RhythmDetect Software System algorithm for providing notifications by identifying rhythms suggestive of atrial fibrillation or atrial flutter events.

ELIGIBILITY:
Inclusion Criteria:

* Adults 22 years of age or older
* Capable of giving informed consent
* U.S. resident
* No prior history of atrial fibrillation or atrial flutter
* Fitbit account, with one of the following devices paired:
* Ionic, Versa, Versa Lite, Versa 2, Versa 3, Charge 3, Charge 4, Inspire HR, Inspire 2, or Sense updated to the latest available firmware.

Exclusion Criteria:

* Diagnosis or history of Atrial Fibrillation at time of consent
* Diagnosis or history of Atrial Flutter at time of consent
* Current use of anticoagulation medication
* Cardiac pacemaker or implantable cardioverter-defibrillator

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450000 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Simultaneous measurement of AF ≥ 30 seconds with detection | 7 days
  Simultaneous measurement of AF ≥ 30 seconds on ECG patch monitor during any of the pulse tachograms that generate the first Irregular Heart Rhythm Detection during ECG monitoring.

SECONDARY OUTCOMES:
Simultaneous measurement of AF ≥ 30 seconds with pulse tachograms | 7 days
  Simultaneous measurement of AF ≥ 30 seconds on the ECG patch monitor during each of the pulse tachograms that contributed to the first Irregular Heart Rhythm Detection, among those detections confirmed by ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lubitz, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - PlushCare, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lubitz SA, McConnell MV, Selvaggi C, Krishnamoorthy A, Atlas SJ, McManus DD, Pagoto S, Singer DE, Pantelopoulos A, Foulkes AS, Faranesh AZ. Wearable Irregular Heart Rhythm Detection Recurrences and Electrocardiographic Atrial Fibrillation Confirmation: The Fitbit Heart Study. Circ Arrhythm Electrophysiol. 2025 Jul;18(7):e013565. doi: 10.1161/CIRCEP.124.013565. Epub 2025 Jun 25. PMID 40557492
- [Derived] Lubitz SA, Faranesh AZ, Selvaggi C, Atlas SJ, McManus DD, Singer DE, Pagoto S, McConnell MV, Pantelopoulos A, Foulkes AS. Detection of Atrial Fibrillation in a Large Population Using Wearable Devices: The Fitbit Heart Study. Circulation. 2022 Nov 8;146(19):1415-1424. doi: 10.1161/CIRCULATIONAHA.122.060291. Epub 2022 Sep 23. PMID 36148649